CLINICAL TRIAL: NCT01377519
Title: Magnetic Resonance-Guided Focused Ultrasound to Treat Uterine Fibroids: A Pilot Randomized, Placebo-Controlled Trial
Brief Title: Magnetic Resonance Guided Focused Ultrasound for Uterine Fibroids
Acronym: PROMISe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2011-06-15; First posted 2011-06-21 (Estimated); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Uterine Fibroids
Keywords: Fibroids; Uterine; Focused Ultrasound; Magnetic Resonance focused ultrasound; HIFU; NOninvasive; Treatment
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MR Guided Focused Ultrasound (Active Comparator)
  Interventions: Procedure: MR Guided Focused Ultrasound
- Placebo MR Guided Focused Ultrasound (Placebo Comparator)
  Interventions: Procedure: Placebo MR Guided Focused Ultrasound

INTERVENTIONS:
Procedure: MR Guided Focused Ultrasound — This is an FDA approved noninvasive treatment for fibroids that uses highly focused ultrasound waves to damage fibroid tissue.
  Arms: MR Guided Focused Ultrasound
Procedure: Placebo MR Guided Focused Ultrasound — This is a placebo treatment that requires a participant to undergo identical procedures as those of the actual MR Guided Focused Ultrasound procedure, but higly focused ultrasound waves are not directed at the uterine fibroid.
  Arms: Placebo MR Guided Focused Ultrasound

SUMMARY:
This is a pilot randomized, blinded, placebo-controlled trial of a noninvasive, FDA approved treatment for uterine fibroids called MR Guided Focused Ultrasound (MRgFUS). Our hypothesis is that MRgFUS provides superior relief of fibroid symptoms compared with the placebo, a sham MRgFUS treatment. The investigators will recruit 20 premenopausal women with symptomatic uterine fibroids to participate in the trial. Participants will be randomly assigned in a 2:1 ratio to the active treatment arm (MRgFUS) versus the sham MRgFUS treatment. Participants will remain blinded to their group assignment for 3 months. After 3 months, participants will be told their treatment group and those assigned to the sham group will be offered complimentary MRgFUS if they desire it. Women will be excluded if they are inappropriate candidates for a 3 month delay in fibroid treatment, such as those with significant anemia. The investigators will assess the change from baseline to 1 and 3 months after treatment in fibroid symptoms, quality of life, fibroid volume measured by MRI, and hematocrit.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Premenopausal
* Symptomatic fibroids
* Fibroids accessible for focused ultrasound treatment

Exclusion criteria:

* Desires future fertility
* Current pregnancy
* Hematocrit <30%
* Emergency room visit in last 3 months for fibroid symptoms
* History of venous thromboembolism
* Fibroids that are: >10cm, non-enhancing with contrast
* Adenomyosis
* Contraindications to undergoing MRI
* Unexplained menstrual irregularity

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Fibroid volume measured on MRI | Change from baseline prior to treatment until 3 months after treatment
Fibroid symptoms reported by participant | Change from baseline prior to treatment to 1 and 3 months after treatment
Red blood cell count (hematocrit) | Change from baseline prior to treatment and 3 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Jacoby, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Jacoby VL, Kohi MP, Poder L, Jacoby A, Lager J, Schembri M, Rieke V, Grady D, Vittinghoff E, Coakley FV. PROMISe trial: a pilot, randomized, placebo-controlled trial of magnetic resonance guided focused ultrasound for uterine fibroids. Fertil Steril. 2016 Mar;105(3):773-780. doi: 10.1016/j.fertnstert.2015.11.014. Epub 2015 Dec 1. PMID 26658133
- See also: Fibroid trials at UCSF — https://clinicaltrials.ucsf.edu/fibroids